CLINICAL TRIAL: NCT00366301
Title: The LANCET Trial: A Randomized Clinical Trial of Lantus for C-reactive Protein Reduction in Early Treatment of Type 2 Diabetes
Brief Title: The LANCET Trial: A Trial of Long-acting Insulin Injection to Reduce C-reactive Protein in Patients With Type 2 Diabetes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Interim analyses demonstrated futility. Thus, recruitment curtailed 10/08.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Aruna Das Pradhan, MD, MPH, Brigham & Women's Hospital, Boston, Massachusetts 02115
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2006-P-000823; Lantus_L_00833
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Results first posted 2010-11-25 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-10

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; insulin; insulin injection; metformin; C-reactive protein; insulin sensitivity; glycemic control; inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Inflammation | interventions — Insulin Glargine; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo pill (Placebo Comparator): Placebo pill
  Interventions: Drug: Placebo pill
- Metformin Pill (Active Comparator): Metformin pill
  Interventions: Drug: metformin
- Insulin Glargine plus placebo pill (Active Comparator): Insulin glargine plus placebo pill
  Interventions: Drug: Insulin glargine injection; Drug: Placebo pill
- Insulin Glargine plus metformin pill (Active Comparator): Insulin Glargine plus metformin pill
  Interventions: Drug: Insulin glargine injection; Drug: metformin

INTERVENTIONS:
Drug: Insulin glargine injection — Once daily for 14 weeks
  Other Names: Lantus
  Arms: Insulin Glargine plus metformin pill; Insulin Glargine plus placebo pill
Drug: metformin — Up to 4 pils per day (2g per day) maximum
  Arms: Insulin Glargine plus metformin pill; Metformin Pill
Drug: Placebo pill — Up to 4 pills per day
  Arms: Insulin Glargine plus placebo pill; Placebo pill

SUMMARY:
The purpose of this study, which is being conducted at 100 centers throughout the United States, is to determine whether Lantus, a long-acting insulin injection, either alone or in combination with metformin, is effective in reducing C-reactive protein (CRP) in adults with type 2 diabetes. CRP is a marker of chronic low-level inflammation, a new risk factor for diabetes, heart attack, stroke, and other cardiovascular events.

DETAILED DESCRIPTION:
Study Rationale

Low-grade systemic inflammation as indicated by elevated levels of C-reactive protein (CRP) is often present in patients with type 2 diabetes. Individuals with type 2 diabetes represent a vulnerable population in which cardiovascular event rates are high and among whom CRP reduction may have the greatest impact. While several classes of oral hypoglycemic agents have been shown to lower CRP, data are not available for newer formulations of long-acting insulins such as Lantus (insulin glargine injection) and no study has comprehensively evaluated the relative merit of insulin-providing versus insulin-sensitizing strategies for this purpose.

Investigational Plan

This is a multicenter, community-based, randomized 2x2 factorial trial of Lantus and metformin among patients with type 2 diabetes treated with either diet or oral monotherapy (other than metformin) only who have poor glycemic control and elevated CRP. The primary endpoint is change in CRP. Secondary endpoints include improvement in insulin sensitivity, glycemic control, blood lipids, as well as selected inflammatory and prothrombotic markers, and adipokine levels.

Limited data suggest that short-term insulin administration in patients with poorly controlled type 2 diabetes may lower CRP, but the benefit of CRP reduction that is unique to insulin therapy and independent of glycemic control per se remains uncertain. The insulin-sensitizing agent metformin, a mainstay of anti-diabetic therapy, has been shown to reduce macrovascular complications among patients with type 2 diabetes and, in some but not all randomized clinical trials, also has a modest CRP-lowering effect. This study is designed to assess whether the use of Lantus either alone or in combination with metformin lowers CRP over a 14-week treatment period.

Eligible men and women age 18 to 79 years with early diabetes on diet only or oral monotherapy with baseline HbA1c 7.0-10% and CRP greater than or equal to 2.0 mg/l will be randomized in a 2X2 factorial fashion as follows. First, participants will be assigned at random to open-label Lantus or no insulin. Then, within these two categories, subjects will be assigned at random to metformin or placebo. Thus, the four resultant treatment groups are Lantus injection and placebo pill, Lantus injection and metformin pill, metformin pill alone, and placebo pill alone. All patients will receive diet and exercise counseling.

This study design will permit testing of the overall effect of Lantus as well as the effect of combination therapy with metformin for CRP reduction at a targeted level of glycemic control (fingerstick fasting blood glucose < 110 mg/dl). All participants will be provided with a glucometer for fingerstick glucose testing calibrated to report plasma-referenced values.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 79
* Type 2 diabetes, treated only by diet or oral drugs other than metformin
* HbA1c greater than or equal to 7% and less than or equal to 10%
* C-reactive protein greater than or equal to 2 mg/L

Exclusion Criteria:

* Baseline use of metformin or insulin
* Type 1 diabetes, history of ketoacidosis or positive anti-GAD antibody
* History of congestive heart failure requiring drug therapy
* Active liver disease
* Kidney impairment
* Recent initiation or change in dose of statins, fibric acid derivatives, angiotensin receptor blockers, nonsteroidal anti-inflammatory agents, or corticosteroids

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2006-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Ridker, MD, MPH, Study Chair — Brigham and Women's Hospital; Aruna Das Pradhan, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Srivastava PK, Pradhan AD, Cook NR, Ridker PM, Everett BM. Randomized Trial of the Effects of Insulin and Metformin on Myocardial Injury and Stress in Diabetes Mellitus: A Post Hoc Exploratory Analysis. J Am Heart Assoc. 2017 Dec 23;6(12):e007268. doi: 10.1161/JAHA.117.007268. PMID 29275373
- [Derived] Pradhan AD, Everett BM, Cook NR, Rifai N, Ridker PM. Effects of initiating insulin and metformin on glycemic control and inflammatory biomarkers among patients with type 2 diabetes: the LANCET randomized trial. JAMA. 2009 Sep 16;302(11):1186-94. doi: 10.1001/jama.2009.1347. PMID 19755697

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at 73 US office-based practices between October 2006 and December 2008.
Pre-assignment Details: Preenrollment evaluation comprised local laboratory testing of hsCRP,HbA1c, and safety parameters (ALT or AST and creatinine). Eligible participants were enrolled in a 2-week run-in. Ability to self-monitor fingerstick blood glucose and perform insulin injection was determined and evaluation for evidence of marked hyperglycemia was undertaken.
Period: Overall Study
Arm/Group | Placebo Pill | Metformin Pill | Insulin Glargine Plus Placebo Pill | Insulin Glargine Plus Metformin Pill
Started | 124 | 126 | 126 | 124
Either 6W or 14W CRP Obtained | 120 | 124 | 124 | 119
Completed | 116 | 120 | 122 | 116
Not Completed | 8 | 6 | 4 | 8
Not completed — Lost to Follow-up | 4 | 4 | 3 | 7
Not completed — Withdrawal by Subject | 4 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Pill | Metformin Pill | Insulin Glargine Plus Placebo Pill | Insulin Glargine Plus Metformin Pill | Total
Number analyzed (Participants) | 124 | 126 | 126 | 124 | 500
Age Continuous [Mean (Standard Deviation); unit: years]
  Mean (SD) | 54.0 (10.9) | 53.8 (11.5) | 53.8 (11.4) | 54.0 (11.7) | 53.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 68 | 83 | 66 | 281
  Male | 60 | 58 | 43 | 58 | 219
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 4 | 19 | 17 | 53
  Not Hispanic or Latino | 110 | 119 | 104 | 105 | 438
  Unknown or Not Reported | 1 | 3 | 3 | 2 | 9
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 91 | 88 | 95 | 91 | 365
  African American | 25 | 34 | 25 | 24 | 108
  Other | 8 | 4 | 6 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage Reduction in C-reactive Protein (CRP)
Time Frame: 14 weeks
Population: As hsCRP was measured at both 6 and 14 weeks, linear mixed models conditioning on baseline hsCRP and adjusting for treatment stratum were constructed with the dependent variable being change in lnCRP. Any subject having either or both 6 week and 14 week measures was included.
Measure: Mean (95% Confidence Interval); unit: Percent CRP Reduction
Arm/Group | Placebo Pill | Metformin Pill | Insulin Glargine Plus Placebo Pill | Insulin Glargine Plus Metformin Pill
Number analyzed (Participants) | 120 | 124 | 124 | 119
Percent CRP Reduction | -19.0 [-27.8 to -9.1] | -16.1 [-25.1 to -6.1] | -2.9 [-13.2 to 8.6] | -20.1 [-28.8 to -10.4]
Statistical Analysis 1: Comparison: Placebo Pill vs Metformin Pill vs Insulin Glargine Plus Placebo Pill vs Insulin Glargine Plus Metformin Pill; As hsCRP was measured at both 6 and 14 weeks, linear mixed models conditioning on baseline hsCRP and adjusting for treatment stratum were constructed with the dependent variable being change in lnCRP. The means at each time point were estimated from a repeated-measures model incorporating all 3 time points. The interventions were assessed by fitting terms corresponding to study drug and treatment arm assignment; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Adjusted models included terms for baseline HbA1c and weight and change in weight at each time point; Percent Change in Log CRP = 20, Standard Error of Mean 10

ADVERSE EVENTS:
Time Frame: 14 weeks
Description: Occurrence of marked hypoglycemia, weight gain, and other adverse events were collected at each of 6 visits.
Arm/Group | Placebo Pill | Metformin Pill | Insulin Glargine Plus Placebo Pill | Insulin Glargine Plus Metformin Pill
Serious Adverse Events (participants affected / at risk) | 3/124 | 8/126 | 2/126 | 0/124
Other Adverse Events (participants affected / at risk) | 12/124 | 18/126 | 21/126 | 17/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Pill (N=124) | Metformin Pill (N=126) | Insulin Glargine Plus Placebo Pill (N=126) | Insulin Glargine Plus Metformin Pill (N=124)
Severe Diarrhea Requiring Hospitalization (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular Tachycardia Requiring Hospitalization (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia Requiring Hospitalization (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis Hospitalization (Infections and infestations) | 1 | 0 (0) | 0 (0) | 0 (0)
Sepsis Hospitazation (Infections and infestations) | 1 (1) | 0 (0) | 0 | 0 (0)
Gastroenteritis Hospitalization (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chest Pain Hospitalization (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Traumatic Injury/Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis Requiring Hospitalization (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Pill (N=124) | Metformin Pill (N=126) | Insulin Glargine Plus Placebo Pill (N=126) | Insulin Glargine Plus Metformin Pill (N=124)
Severe Hypoglycemia (Endocrine disorders) | 1 (1) | 3 (3) | 3 (3) | 6 (6) — Subjects were queried at each study visit.
Hyperglycemia: Confirmed Fasting Glucose >= 250 mg/dl (Endocrine disorders) | 10 (10) | 1 (1) | 4 (4) | 1 (1)
Hyperglycemia: Any Self-Monitor Blood Glucose >= 400 mg/dl (Endocrine disorders) | 3 (3) | 0 (0) | 3 (3) | 1 (1)
Weight Gain >= 5% of Baseline (Endocrine disorders) | 3 (3) | 4 (4) | 14 (14) | 8 (8)
Gastrointestinal Adverse Event (e.g. diarrhea not requiring hospitalization) (Gastrointestinal disorders) | 3 (3) | 13 (13) | 4 (4) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No